CLINICAL TRIAL: NCT04554186
Title: Ultrasound Guided Serratus Anterior Plane Block Versus Thoracic Paravertebral Block in Emergency Department Rib Fracture
Brief Title: Serratus Anterior Plane Block Versus Thoracic Paravertebral Block.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Shehata, Assistant lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112-11/2018
Record Dates: First submitted 2020-09-12; First posted 2020-09-18 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Rib Fractures; Analgesia
Keywords: Fracture rib; TPVB; SAPB
MeSH Terms: conditions — Rib Fractures; Agnosia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Serratus anterior plane block (Experimental): 20 patients will receive SAP block with 0.4 ml / kg bupivacaine 0.125% then continuous infusion through a catheter at rate of 7 ml / hour to max 10 ml / hour of bupivacaine 0.0625%
  Interventions: Procedure: Serratus anterior plane block
- Thoracic Paravertebral block (Active Comparator): 20 patients will receive TPVB 0.4ml / kg bupivacaine 0.125% then continuous infusion through a catheter at rate of 7 ml / hour to max 10 ml / hour of bupivacaine 0.0625%
  Interventions: Procedure: Thoracic Paravertebral block
- Control group (Placebo Comparator): 20 patients will receive Fentanyl patch 50 microgram
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Serratus anterior plane block — Injection of bupivacaine between serratus anterior plane and latissimus dorsi muscle using ultrasound
  Arms: Serratus anterior plane block
Procedure: Thoracic Paravertebral block — Injection of bupivacaine in the thoracic Paravertebral space using ultrasound
  Arms: Thoracic Paravertebral block
Procedure: Control — Place a fentanyl patch 50 microgram
  Arms: Control group

SUMMARY:
Compare between serratus anterior plane block and thoracic Paravertebral block in analgesia for patients with multiple rib fractures

DETAILED DESCRIPTION:
The study will be conducted in a prospective randomised controlled. Patients will be allocated into three groups

Control group:

The patient will receive fentanyl patch 50 microgram

TPVB group:

The patient will receive thoracic vertebral plane lock 0.4ml/kg bupivacaine 0.1 25% will be administered. For continuous infusion catheter will be inserted . Then a rate of 7ml / hour to max 10 ml / hour of bupivacaine 0.0625%

SAPB group,:

Patient will receive serratus anterior plane block 0.4ml / kg bupivacaine 0.125% will be injected to open the space then a catheter will be advanced For continuous infusion of 0.0625 % bupivacaine at 7 ml / hour

ELIGIBILITY:
Inclusion Criteria:

* ASA 1_3 Age 18_60 Unilateral fracture ribs

Exclusion Criteria:

* Drug allergy Morbid obese Opioid dependence Patients refuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
VAS score | 24 hour
  Visual analogue pain score describe by the patient

SECONDARY OUTCOMES:
Total analgesic consumption | 24 hour
  Total opioid consume by the patient in 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Amany K Aboelhassan, Study Chair — Minia University Hospital
Locations (1):
- Minia university hospital, Minya, Egypt